CLINICAL TRIAL: NCT03991728
Title: International, Multicenter, Prospective Registry to Collect Data of Patients Treated With Alloplastic Total Temporomandibular Joint (TMJ) Replacements
Brief Title: Alloplastic Total Temporomandibular Joint (TMJ) Replacement Registry
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: TMJ Replacement
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular joint; TMJ replacement; Trauma; Ankylosis; Degenerative joint disease; Registry
MeSH Terms: conditions — Temporomandibular Joint Disorders; Wounds and Injuries; Ankylosis; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alloplastic total TMJ replacement: All treatments will remain the standard (routine) care procedures based on individual clinician's judgment and the patient characteristics. The registry does not dictate any specific treatment.

SUMMARY:
Prospective data will be collected in approximately 200 patients treated with an TMJ replacement. Patients will be followed up according to the standard (routine) for up to 5 years after the treatment. Data collection will include underlying disease, treatment details, functional and patient reported outcomes (PRO)s and anticipated or procedure-related adverse events (i.e. complications).

This registry is designed to be able to assess the number of patients who refuse alloplastic total TMJ replacement. Therefore, the participating sites are asked to register all cases of refused TMJ replacements too.

DETAILED DESCRIPTION:
More in detail this registry has the following objectives:

* To describe clinical indications for TMJ replacement, and treatment patterns (including differences among regions if feasible)
* To describe the clinical evolution and outcomes of patients treated with a TMJ replacement
* To explore the relationship(s) between treatment, outcome(s) and quality of life (QoL).
* To identify predictive factors for favorable outcomes (pain reduction, range of motion (ROM), occlusal status, QoL) in patients treated with TMJ replacement.
* To describe the reasons of patients who refused TMJ replacements

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and or older
* Patients requiring alloplastic total TMJ replacement
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/informed consent form (ICF)
  * Willingness and ability to participate in the registry according to the Registry Plan (RP)
  * Signed and dated ethics committee (EC) / Institutional review board (IRB) approved written informed consent

Exclusion Criteria:

* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the study period
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring alloplastic total TMJ replacement
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2032-09 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
The registry has no primary but several objectives. | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  due to the study design, no primary objective has been defined and therefore no primary outcome measure either

SECONDARY OUTCOMES:
Demographics | pre-operative
  Year of birth Gender Smoking
Comorbidities | pre-operative
  Concomitant diseases will be assessed using the Charlson Comorbidity Index (CCI). This score assesses the comorbidity level by considering both the number and severity of pre-defined comorbid conditions. It provides a weighted score of a patient's comorbidities which can be used to predict mortality rates
Refusal of alloplastic total TMJ replacement surgery | pre-operative
  For patients who require alloplastic total TMJ replacement but refuse surgery, the reason(s) for refusal will be collected.
Clinical and functional outcomes - Mandibular movements | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  Interincisial opening/maximal opening Lateral movements Protrusive movement
Clinical and functional outcomes - Occlusal status | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  Occlusion will be assessed according to Angle's classification:
Clinical and functional outcomes - Dentition | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  Dental status will be recorded as:
  * Edentulous
  * Complete dentition
  * Partial dentition In case of partial dentition, missing teeth will be recorded individually using the Fédération Dentaire Internationale (FDI) tooth numbering formula .
Clinical and functional outcomes - Helkimo Clinical dysfunction index | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  The dysfunction of the mandible will be evaluated by means of the Helkimo index. The Helkimo index is based on the assessment of five different symptoms.
Patient Reported Outcomes - Pain numeric rating scale (NRS) | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  The Pain NRS is an 11-point scale where the end points are the extremes of no pain (0 points), to worst imaginable pain (10 points). It measures subjective intensity of pain and the patient rates his/her overall or average daily pain.
  Will be assessed independently for each site.
Patient Reported Outcomes - Jaw function NRS | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  The jaw function NRS is an 11-point scale where the end points are the extremes of normal jaw movement (0 points), to no jaw movement (10 points). It measures subjective jaw function.
Patient Reported Outcomes - Diet limitation NRS | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  The diet limitation NRS is an 11-point scale where the end points are the extremes of no restrictions (0 points), to liquids only (10 points). It measures subjective diet limitations.
Patient Reported Outcomes - EuroQoL five dimension (EQ-5D-5L) | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months
  The EQ-5D-5L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Patient Reported Outcomes - Oral Health Impact Profile (OHIP) - 14 | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months
  The OHIP is concerned with impairment and three functional status dimensions (social, psychological and physical) which represent four of the seven quality of life dimensions proposed by Patrick and Bergner. Hence, it excludes perceptions of satisfaction with oral health, changes in oral health, prognosis or self-reported diagnoses. Furthermore, the OHIP aims to capture impacts that are related to oral conditions in general, rather than impacts that may be attributed to specific oral disorders or syndromes. All impacts in the OHIP are conceptualized as adverse outcomes, and therefore the instrument does not measure any positive aspects of oral health. The OHIP consists of 14 items evaluated using a 5-point Likert from "Never" to "Very often " in which higher scores indicated worse outcomes. It has validated translations to Swedish, Spanish, German, Hindi and further more.
Anticipated treatment or condition-related adverse events (i.e. complications) | from the pre-operative assessment until 60 months after surgery (10 days / 3 months / 6 months / 12 months / 24 months / 60 months)
  In this registry, only anticipated condition, treatment-, or implant-related adverse events (i.e. complications) will be documented in the electronic case report form (eCRF) from the time of consent onwards.
  In the context of the registry, these events are considered as events of scientific interest, i.e. events that can clearly be connected to the treatment(s) or the medical condition under investigation. These events do not require immediate reporting unless they occur at a higher frequency and/or severity to that cited in the literature
Survival | 10 days / 3 months / 6 months / 12 months / 24 months / 60 months
  Follow up (FU) visits will be scheduled and performed according to the local standard of care and at each scheduled visit the patient's survival will be documented. In case a patient misses a scheduled visit, it will be assessed if the patient is still alive, which can be done via phone call.
Radiological parameters - Displacement of ramus component | pre-operative / 10 days / 12 months / 24 months
  All images (preferably computed tomography (CT) / cone beam (CB) CT scan) taken as part of the standard (routine) will be collected and 'displacement of ramus component' evaluated by local investigator:
Radiological parameters - Fracture of ramus component | pre-operative / 10 days / 12 months / 24 months
  All images (preferably computed tomography (CT) / cone beam (CB) CT scan) taken as part of the standard (routine) will be collected and evaluated by local investigator if a 'fracture of the ramus component' occurred
Radiological parameters - Screw loosening | pre-operative / 10 days / 12 months / 24 months
  All images (preferably computed tomography (CT) / cone beam (CB) CT scan) taken as part of the standard (routine) will be collected and evaluated by local investigator if 'screw loosening' occurred
Radiological parameters - Resorption/ osteolysis of surrounding bone | pre-operative / 10 days / 12 months / 24 months
  All images (preferably computed tomography (CT) / cone beam (CB) CT scan) taken as part of the standard (routine) will be collected and 'resorption/ osteolysis of surrounding bone' evaluated by local investigator
Radiological parameters - Status of bone grafts if used (displaced/ resorbed/ healed) | pre-operative / 10 days / 12 months / 24 months
  All images (preferably computed tomography (CT) / cone beam (CB) CT scan) taken as part of the standard (routine) will be collected and 'status of bone grafts if used (displaced/ resorbed/ healed)' evaluated by local investigator
Radiological parameters - Presence of ectopic bone | pre-operative / 10 days / 12 months / 24 months
  All images (preferably computed tomography (CT) / cone beam (CB) CT scan) taken as part of the standard (routine) will be collected and 'presence of ectopic bone' evaluated by local investigator

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Thor, MD, Principal Investigator — Oral and Maxillofacial surgery Uppsala University Hospital; Vinay V Kumar, MD, Principal Investigator — Oral and Maxillofacial surgery Uppsala University Hospital
Locations (23):
- Hospital BP - A Beneficência Portuguesa de São Paulo, São Paulo, Brazil
- Estetica Maxilofacial, Bogotá, Colombia
- Rigshospitalet, Copenhagen, Denmark
- Germany (4):
  - Hannover Medical School, Hanover
  - University Hospital Leipzig, Leipzig
  - Klinikum der Johannes Gutenberg Universität Mainz, Mainz
  - Klinikum der LMU München, Munich
- India (2):
  - Sri Shankara Cancer Hospital and Research Center, Bangalore
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- New Zealand (2):
  - Waikato DHB, Christchurch
  - Hutt Hospital, Lower Hutt
- Mayo Hospital, Lahore, Pakistan
- Wojewódzki Specjalistyczny Szpital Dziecięcy, Olsztyn, Poland
- National Medical and Surgical Center named after N.I. Pirogov" of the Ministry of Healthcare of the Russian Federation, Moscow, Russia
- Clinic for Maxillofacial Surgery, University of Belgrade, Belgrade, Serbia
- King Edward VIII Hospital, Durban, South Africa
- 12 de Octubre University Hospital, Madrid, Spain
- Sweden (4):
  - Falu Hospital, Falun
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No